CLINICAL TRIAL: NCT00503841
Title: A Pilot Study of the Effect of Erlotinib (Tarceva®) on Biomarkers in Estrogen Receptor Negative Breast Cancer Expressing the Epidermal Growth Factor Receptor and Interleukin 1α
Brief Title: Erlotinib in Treating Women Undergoing Surgery For Stage I, Stage II, or Stage III Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All enrolled participants were screen failures, no data were collected for outcome measures.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elaina Gartner, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000554965; P30CA022453 (NIH); WSU-2006-138; NCT01654757 (obsolete NCT alias)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; recurrent breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Erlotinib Hydrochloride; Immunohistochemistry; Biopsy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- erlotinib hydrochloride (Experimental): Patients receive erlotinib hydrochloride PO (orally) QD (every day) on days -14-0 immediately prior to scheduled surgery. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: biopsy; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Drug: erlotinib hydrochloride — Patients receive erlotinib hydrochloride PO (orally) QD (every day) on days -14-0 immediately prior to scheduled surgery. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Other Names: CP-358,774; Erlotinib; OSI-774; Tarceva
Other: immunohistochemistry staining method — Assessed at the time of the initial biopsy and at the time of surgery.
Other: laboratory biomarker analysis — Correlative studies
Procedure: biopsy — 14 days prior to surgery
Procedure: conventional surgery — 14 days after taking study drug erlotinib hydrochloride.
Procedure: neoadjuvant therapy — 14 days after taking study drug erlotinib hydrochloride.

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This clinical trial is studying how well erlotinib works in treating women undergoing surgery for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the effect of erlotinib hydrochloride on expression of interleukin (IL)-1α in patients with estrogen receptor (ER-)-negative, EGFR-positive and IL-1α-positive breast cancer.

Secondary

* To estimate the effect of erlotinib hydrochloride on expression of nuclear NF-κB and amphiregulin (AR) in patients with ER-negative, EGFR-positive and IL-1α-positive breast cancer.
* To estimate the effect of erlotinib on tumor cell proliferation (Ki67) and apoptosis (TUNEL).
* To estimate the rates of IL-1α, nuclear NF-κB, and AR expression in patients with ER-negative, EGFR-positive breast cancer.
* To follow the clinical course of patients with resectable ER-negative, EGFR-positive and IL-1α-positive breast cancer.
* To assess the toxicity of a 15-day regimen of daily oral administration of erlotinib hydrochloride in participants with ER-negative, EGFR-positive and IL-1α-positive breast cancer.

OUTLINE: This is an open-label, pilot study. Patients are stratified according to HER2 status (positive vs negative).

Patients receive oral erlotinib hydrochloride once daily on days -14 to 0 in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery on day 0.

Tissue samples are collected at baseline and examined for expression of estrogen receptor, progesterone receptor, HER2, EGFR, interleukin (IL)-1α, amphiregulin, and NF-kB. Tissue samples collected at surgery are examined for IL-1α, NF-kB, and amphiregulin by IHC.

Following surgery, patients will be contacted 1 week post-surgery (± 1 day) or 1 week post-withdrawal from study (± 1 day) by phone call or clinic visit to assess toxicity. After that, patients will be followed and treated according to standard of care practices. If patients choose to follow-up with an oncologist outside of our institution, they or their oncologist will be contacted every 6 months for updated information on their conditions.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion

* Cytologically or histologically confirmed adenocarcinoma of the breast

  * Stage I-III disease
  * BI-RADS 4 or 5 abnormalities on breast imaging and undergoing core needle biopsy for diagnosis
  * Participants must have a lesion of at least 1-cm on breast imaging studies (mammogram, ultrasound, or MRI)
  * Participants must have breast cancer amenable to surgery with curative intent and must have agreed to undergo such surgery

    * The surgical procedure must be scheduled in the near future to accommodate a treatment period of no less and no more than 15 days
* Clinically positive for the overexpression of EGFR and interleukin-1α
* Clinically negative for expression of the estrogen receptor (ER-negative) and progesterone receptor (PgR-negative)

  * May be positive or negative for HER2

Exclusion

* Locally advanced or metastatic disease not amenable to surgery
* Known brain metastases

PATIENT CHARACTERISTICS:

Inclusion

* Female
* Menopausal status not specified
* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* ANC ≥ 1000/mm³
* Platelet count ≥ 75,000/mm³
* AST and ALT ≤ 2.5 times upper limits of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 2 times ULN
* Hemoglobin > 9 g/dL
* Creatinine within normal institutional limits OR creatinine clearance >60 mL/min
* Negative serum pregnancy test within 7 days of enrollment for pre-menopausal women and women within 6 months of menopause
* Women of child-bearing potential and their partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

Exclusion

* Pregnant or nursing
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib hydrochloride
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

Exclusion

* Received any other therapy (i.e., surgery, radiation, hormone treatment, biologic therapy, and/or chemotherapy) for the treatment of breast cancer
* Concurrent use of anti-neoplastic or anti-tumor agents not part of the study therapy, including chemotherapy, radiation therapy, immunotherapy, and hormonal anticancer therapy
* Receiving any other investigational agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaina M. Gartner, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 participants signed consent starting 1-9-08 and recruitment ending with the last participant signing on 1-19-10. All participants enrolled onto screening portion of study, but none were ever put onto the "treatment" portion of the study.
Pre-assignment Details: All participants that signed consent were screen failures.
Groups:
- Erlotinib Hydrochloride: If participants would have went onto study they would receive erlotinib(Tarceva®)hydrochloride 150 mg/day starting dose PO (orally) self-administered, QD (every day) on days -14 until day 0 immediately prior to scheduled surgery, Tissue sent for biomarker modulation analysis
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Biomarker analysis performed, toxicity monitored for 7 days following last dose of erlotinib (Tarceva®)
Period: Overall Study
Arm/Group | Erlotinib Hydrochloride
Started | 44
Completed | 0
Not Completed | 44
Not completed — All screen failures | 44

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib Hydrochloride: If participants would have went onto study they would receive erlotinib hydrochloride PO (orally) QD (every day) on days -14-0 immediately prior to scheduled surgery. Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 52 [24 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Effect of Erlotinib Hydrochloride on Expression of IL-1a in Patients With ER- Negative, EGFR- Positive and (IL-)1a-positive Breast Cancer
Time Frame: Baseline and day 0
Population: No participants received the study drug erlotinib hydrochloride.
Groups:
- Erlotinib Hydrochloride: Patients must be willing to consider treatment with erlotinib, in the event they are eligible for the treatment phase of the study. Erlotinib (Tarceva®) will be self-administered in an open-label, unblinded manner to all patients enrolled in the study. During the treatment period, patients will receive single-agent erlotinib (Tarceva®), at a dose of 150 mg/day mg by mouth. Patients will be instructed to take tablets once daily. The day of planned surgical resection of the invasive breast cancer will be considered day 0. Patients will undergo baseline physical examination and performance status evaluation on or before day -14. Patients will begin treatment with erlotinib 150 mg (1 tablet) orally daily on day -14 and it will be continued for a total of 15 days, through day 0.
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 0

2. Secondary Outcome: Effect of Erlotinib Hydrochloride on Expression of NF-κB and AR in Patients With ER-negative, EGFR-positive and IL-1a-positive Breast Cancer
Time Frame: Baseline and day 0
Population: No data collected for secondary hypotheses.
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 0

3. Secondary Outcome: Effect of Erlotinib Hydrochloride on Tumor Cell Proliferation (Ki67) and Apoptosis (TUNEL)
Time Frame: Baseline and day 0
Population: No data collected for secondary hypotheses.
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity of a 15-day Regimen of Daily Oral Administration of Erlotinib Hydrochloride
Time Frame: At day -7, prior to surgery, and 1 week post-surgery
Population: No data collected for secondary hypotheses.
Arm/Group | Erlotinib Hydrochloride
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No patients were actually treated on the study.
Groups:
- Erlotinib Hydrochloride: Patients will be instructed to take tablets once daily.Patients will begin treatment with erlotinib 150 mg (1 tablet) orally daily on day -14 and it will be continued for a total of 15 days, through day 0.The day of planned surgical resection of the invasive breast cancer will be considered day 0.
Arm/Group | Erlotinib Hydrochloride
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
All 44 participants that signed consent were screen failures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No